CLINICAL TRIAL: NCT06284174
Title: Effectiveness of Povidone-Iodine Versus Chlorhexidine Gluconate Solutions in Reducing Microbial Contamination in Spinal Surgery Wounds During Intraoperative Soaking.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: B-BR-109-054-T
Record Dates: First submitted 2024-02-21; First posted 2024-02-28 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Spine Infection
Keywords: Spine surgery, Providine-iodine, Chlorohexidine gluconate, surgical wound infection
MeSH Terms: conditions — Surgical Wound Infection | interventions — chlorhexidine gluconate

STUDY DESIGN:
Intervention Model Description: This research will include patients diagnosed with lumbar spinal stenosis causing nerve compression, who are scheduled for open spinal decompression and fusion surgery. Patients will be randomly assigned to one of three groups: a control group (soaked with 0.9% normal saline), an iodine group (soaked with 3.5% povidone-iodine solution), and a CHG group (soaked with 0.05% chlorhexidine gluconate). All groups will receive the same surgical pre-care, preoperative disinfection, and prophylactic antibiotics. Before wound closure, each group will undergo different irrigation solutions for soaking the wound for three minutes followed by rinsing with copious saline. Samples from deep and superficial tissues and implants will be taken for bacterial culture and molecular biochip analysis.
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients will be randomly assigned by computer to one of three groups: a control group (soaked with 0.9% normal saline), an iodine group (soaked with 3.5% povidone-iodine solution), and a CHG group (soaked with 0.05% chlorhexidine gluconate). All groups will receive the same surgical pre-care, preoperative disinfection, and prophylactic antibiotics.
  All patients understood the experimental process and signed the consent form. The patients did not know the group they were assigned to during the whole process. The bacterial culturers, examiners and clinical outcome assessors did not know the patient group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- control group (Placebo Comparator): Before wound closure, patients will undergo 0.9% normal saline irrigation solutions for soaking the wound for three minutes followed by rinsing with copious saline.
  Interventions: Drug: Povidone-iodine solution; chlorhexidine gluconate
- povidone-iodine group (Experimental): Before wound closure, patients will undergo 3.5% povidone-iodine solutions for soaking the wound for three minutes followed by rinsing with copious saline.
  Interventions: Drug: Povidone-iodine solution; chlorhexidine gluconate
- CHG group (Experimental): Before wound closure, patients will undergo 0.05% chlorhexidine gluconate (CHG) solution for soaking the wound for three minutes followed by rinsing with copious saline.
  Interventions: Drug: Povidone-iodine solution; chlorhexidine gluconate

INTERVENTIONS:
Drug: Povidone-iodine solution; chlorhexidine gluconate — Before wound closure, each group will undergo different irrigation solutions for soaking the wound for three minutes followed by rinsing with copious saline.

SUMMARY:
This study aims to assess the efficacy of intraoperative wound irrigation with iodine-containing and chlorhexidine-containing solutions in reducing bacterial colonization during spine surgery, and to determine which solution is more effective. Additionally, we aim to evaluate any side effects associated with the use of these two antiseptic solutions for wound irrigation.

DETAILED DESCRIPTION:
Study Background: Infection is a challenging complication in spinal surgery, with various methods proposed to reduce intraoperative bacterial load and subsequently lower postoperative infection rates. The use of iodine-containing solutions on surgical wounds has been shown to effectively reduce infection rates after spinal surgery. However, some studies suggest that iodine solutions may impair fibroblast activity, affecting wound healing. Chlorhexidine is another effective antimicrobial agent, which, compared to iodine solutions, has similar antimicrobial efficacy without hindering wound recovery. Its use for intraoperative irrigation in joint replacement surgery has been reported to effectively reduce postoperative infections. Yet, evidence of its effectiveness as an irrigation solution in spine surgery is lacking, and previous studies have rarely focused on intraoperative wound sampling to investigate whether irrigation solutions can effectively reduce microbial residue.

Study Objective: The aim of this experiment is to evaluate whether the use of iodine-containing solutions and chlorhexidine for wound irrigation before closing spinal surgery wounds can effectively reduce the positive rate of bacterial cultures, and to assess which has stronger functionality and any associated side effects.

Study Methods: This research will include patients diagnosed with lumbar spinal stenosis causing nerve compression, who are scheduled for open spinal decompression and fusion surgery. Patients will be randomly assigned to one of three groups: a control group (soaked with 0.9% normal saline), an iodine group (soaked with 3.5% povidone-iodine solution), and a CHG group (soaked with 0.05% chlorhexidine gluconate). All groups will receive the same surgical pre-care, preoperative disinfection, and prophylactic antibiotics. Before wound closure, each group will undergo different irrigation solutions for soaking the wound for three minutes followed by rinsing with copious saline. Samples from deep and superficial tissues and implants will be taken for bacterial culture and molecular biochip analysis.

Study Significance: Infections in spinal surgery have a significant impact on patient outcomes and healthcare costs. This study aims to confirm whether pre-wound closure soaking with antimicrobial solutions can effectively reduce bacterial load inside and outside the wound to lower the risk of postoperative infection.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were diagnosed with lumbar spinal stenosis need to undergo posterior lumbar decompression with fusion surgery.

Exclusion Criteria:

* People who are allergic to disinfectants (Providine or CHG)
* The surgical site has been operated before.
* Patients under active infection status.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Bacteria culture and Polymerase chain reaction exam | one week postoperatively.
  Samples from deep and superficial tissues and implants will be taken for bacterial culture and PCR analysis. Positive means bacterial growth.

SECONDARY OUTCOMES:
Post operative infection | within 6 months after surgery
  Patient develops symptomatic wound infection will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
Can share de-identified data